CLINICAL TRIAL: NCT02205918
Title: Integrative Examination of Neurobehavioral Mechanisms in Tic Suppression
Brief Title: Brain-Behavior Interactions in Tic Suppression
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2017-25550
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Tourette's Syndrome; Chronic Motor Tic Disorder; Chronic Vocal Tic Disorder
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sham TMS: Participants in this group will receive one, 30 minute session of inactive ("sham") TMS.
  Interventions: Other: Sham TMS
- Active TMS: Participants in this group will receive one, 30 minute session of 1hz TMS.
  Interventions: Other: Active TMS

INTERVENTIONS:
Other: Active TMS — There will be one, 30-minute TMS session. Participants randomly assigned to this group will receive 1hz "active" TMS. Tics and urges will be monitored immediately before and after TMS.
  Groups: Active TMS
Other: Sham TMS — There will be one, 30-minute TMS session. Participants randomly assigned to this group will receive inactive ("sham") TMS. Tics and urges will be monitored immediately before and after TMS.
  Groups: Sham TMS

SUMMARY:
The purpose of this study is to examine how the brain and environment interact to influence children's ability to suppress tics using a medical technology called Transcranial Magnetic Stimulation (TMS).

DETAILED DESCRIPTION:
Objectives: This study will recruit youth with chronic tics. Chronic tics are the most common movement disorder in children. The goal of the study is to learn how the brain and environment influence children's ability to suppress tics. Specifically, we want to learn how tics are influenced by a certain part of the brain called the supplementary motor area (SMA). This part of the brain is thought to be more active in people with tics. This will be the first study to look at the relationship between SMA, tic suppression, and urges to tic.

Research Procedures: The study will take place over the course of three days within a week (about 5 hours total). The study will examine the relationship between the SMA and tic suppression using a non-invasive medical technology called Transcranial Magnetic Stimulation (TMS). Participants will have a diagnostic interview, MRI brain scan (used to find the location of the SMA), and TMS. Participants will be asked to try to suppress tics before and after TMS. The information that will be collected from participation includes information about tic symptoms, emotional and behavioral functioning, and brain activity (from MRI brain images and TMS results).

ELIGIBILITY:
Inclusion Criteria:

* Presence of motor and/or vocal tics for at least one year
* English fluency

Exclusion Criteria:

* Participants with medical conditions that are contraindicated for TMS (history of any known intracranial pathology, epilepsy or seizures, traumatic brain injury, brain tumor, stroke, implanted medical devices, current pregnancy or girls of childbearing age not using effective contraception, or any other serious medical conditions
* Left-handedness
* Previous diagnosis of psychosis, autism spectrum disorder, mental retardation, or cognitive disability
* Inability to undergo MRI
* Substance abuse or dependence within the past year
* History of ≥3 sessions of Habit Reversal Therapy or other treatment primarily comprised of tic suppression strategies
* Current suicidal intent
* Current neuroleptic medications, as these medications are known to lower seizure threshold

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Tic frequency | Day 3
  Tics will be observed and counted

SECONDARY OUTCOMES:
Urge to tic | Day 3
  The participant will be asked to give subjective ratings of premonitory urge intensity

CONTACTS AND LOCATIONS:
Overall Officials: Christine Conelea, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No